CLINICAL TRIAL: NCT05641675
Title: Feasibility Study to Determine if Novel Wearable Monitoring System and Machine-Learning Algorithm Can Model Continuous Pulmonary Artery Pressure Recordings in Human Subjects
Brief Title: Non-invasive Pulmonary Artery Prediction (ADOPTS)
Acronym: ADOPTS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Silverleaf Medical Sciences INC (Industry)
Collaborators: VA Loma Linda Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: ADOPTS_VALL
Record Dates: First submitted 2022-11-29; First posted 2022-12-08 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-11

CONDITIONS: Heart Failure; Pulmonary Arterial Hypertension
Keywords: Pulmonary artery pressure; Electrocardiogram; Heart failure; Machine Learning
MeSH Terms: conditions — Heart Failure; Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- right heart catheterization cohort: The study investigators will screen up to 50 Veterans undergoing right heart catheterization for clinical indications with the intention to consent up to 20 Veterans. Veterans will be screened by study investigators. Veterans who decline to consent and vulnerable populations (pregnant, incapacitated, incarcerated) will be excluded from the study.
  Interventions: Diagnostic Test: right heart catheterization

INTERVENTIONS:
Diagnostic Test: right heart catheterization — Connect to a heart monitor to record heart rate, blood pressure and blood oxygen levels Place sterile sheets on chest and neck (or groin area) Clean the skin over the neck or groin Give local anaesthetic to numb the area (this may sting a little when it is given) Gently pass a catheter into a vein to the heart Record pressure readings from the heart chambers and lungs Give medication, depending on heart's pressure readings Remove the catheter and apply pressure where it was inserted

SUMMARY:
A proprietary machine-learning algorithm has been developed to model continuous pulmonary artery pressure (PAP), a physiologic marker of cardiopulmonary function. The algorithm was developed from PAP recordings obtained during invasive right heart catheterization. The study will evaluate whether this algorithm can perform as well when embedded into a non-invasive wearable device that records EKG, heart sounds, and thoracic impedance has yet to be established.

DETAILED DESCRIPTION:
A prototype device will be supplied by Silverleaf Medical Science (Redlands, CA) to record these signals. This study will take place at Loma Linda VA, in the cardiac catheterization lab as an add-on to clinically-indicated right heart catheterizations, and under the supervision of heart failure and interventional cardiologists. The investigators will screen and enroll 20 Veterans who consent to participate in the study. Veterans who decline to consent and vulnerable populations will be excluded from the study. The investigators will obtain simultaneous recordings from the prototype device (EKG, heart sounds, and thoracic impedance) and from the PAP catheter , both at rest (5 minutes), and in response to physiological maneuvers: hand grip, passive leg raise, and Valsalva (1 minute recordings with 1-minute breaks). De-identified recordings from the prototype device will be shared with the team at Silverleaf Medical Science to derive a computed PAP. The investigators will test the hypothesis that computed PAP is no different than measured PAP. If the algorithm can produce a computed PAP with high accuracy,'[it would be the first wearable system to non-invasively report PAP.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and authorization to use and disclose health information.
* 20 years of age or older.
* Diagnosis of HF for >3 months, with preserved or reduced left ventricular ejection fraction (LVEF).
* Female subjects of childbearing age with a negative urine or serum pregnancy test at the time of the right heart cauterization procedure and trial.

Exclusion Criteria:

* Active infection.
* Unable to tolerate a right heart catheterization (RHC), in the investigator's opinion.
* Implantation of cardiac resynchronization therapy (CRT)<3 months before enrollment.
* Enrolled in concurrent studies that may confound the results of this study.
* Clinical condition that would not allow them to complete the study, in the investigator's opinion.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study investigators will screen up to 50 Veterans undergoing right heart catheterization for clinical indications with the intention to consent up to 20 Veterans. Veterans will be screened by study investigators. Veterans who decline to consent and vulnerable populations (pregnant, incapacitated, incarcerated) will be excluded from the study.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Major Outcome | the Swan-Ganz catheter obtains the pulmonary artery pressures for a minimum of 5 minutes
  The primary outcome of this study is to determine if a machine-learning algorithm with data from a wearable device can reproduce simultaneous PAP measurement obtained during right heart catheterization.

CONTACTS AND LOCATIONS:
Overall Officials: Jay Patel, Principal Investigator — Loma Linda Veterans Administration Healthcare System; Islam Abudayyeh, Study Director — Silverleaf Medical Sciences INC; Jianwei Zheng, Ph.D., Study Chair — Silverleaf Medical Sciences INC
Locations (1):
- Loma Linda Veterans Administration Healthcare System, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Zheng J, Abudayyeh I, Mladenov G, Struppa D, Fu G, Chu H, Rakovski C. An artificial intelligence-based noninvasive solution to estimate pulmonary artery pressure. Front Cardiovasc Med. 2022 Aug 24;9:855356. doi: 10.3389/fcvm.2022.855356. eCollection 2022. PMID 36093166